CLINICAL TRIAL: NCT00000507
Title: Intravenous Streptokinase in Acute Myocardial Infarction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 26; R01HL030300 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 1994-10

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction; Myocardial Ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction; Myocardial Ischemia | interventions — Streptokinase

INTERVENTIONS:
Drug: streptokinase

SUMMARY:
To determine whether the administration of intravenous streptokinase (SK) early in the course of acute, transmural myocardial infarction would limit myocardial damage.

DETAILED DESCRIPTION:
BACKGROUND:

Determination of the potential value of thrombolytic therapy in patients with acute myocardial infarction was an issue of major importance in 1983. An estimated 1.4 million heart attacks occurred each year, of which over 500,000 were fatal. Reduction of mortality required an effective means to reduce infarct size. Studies indicated that reperfusion represented a potent means of achieving salvage of ischemic myocardium. Pilot clinical studies indicated that reperfusion could be achieved in a substantial percentage of patients by lysis of coronary thrombosis with both intracoronary and intravenous streptokinase administration. Intracoronary thrombolysis was receiving widespread clinical applications but had many limitations. The intracoronary route took 90-120 minutes longer to administer than the intravenous route. Because intracoronary therapy required the availability of a catheterization laboratories and highly skilled invasive cardiologists, this treatment was not available to large numbers of patients who were hospitalized in smaller community hospitals.

DESIGN NARRATIVE:

Randomized design with two groups and fixed sample size. Control patients received routine coronary care. The treatment group received intravenous streptokinase plus conventional care. This was followed with intravenous heparin and warfarin. The primary endpoint was 14 day mortality. Secondary endpoints included angiographic patency of the involved coronary artery at 10 to 14 days, left ventricular function, segmental wall motion analysis, and myocardial infarction size at 30-45 days.

ELIGIBILITY:
Men and women, aged less than 75. Myocardial infarction onset within six hours.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1983-08; Study Completion 1994-10

REFERENCES:
- [Background] Martin GV, Sheehan FH, Stadius M, Maynard C, Davis KB, Ritchie JL, Kennedy JW. Intravenous streptokinase for acute myocardial infarction. Effects on global and regional systolic function. Circulation. 1988 Aug;78(2):258-66. doi: 10.1161/01.cir.78.2.258. PMID 3396164
- [Background] Ritchie JL, Cerqueira M, Maynard C, Davis K, Kennedy JW. Ventricular function and infarct size: the Western Washington Intravenous Streptokinase in Myocardial Infarction Trial. J Am Coll Cardiol. 1988 Apr;11(4):689-97. doi: 10.1016/0735-1097(88)90197-0. PMID 3280640
- [Background] Kennedy JW, Martin GV, Davis KB, Maynard C, Stadius M, Sheehan FH, Ritchie JL. The Western Washington Intravenous Streptokinase in Acute Myocardial Infarction Randomized Trial. Circulation. 1988 Feb;77(2):345-52. doi: 10.1161/01.cir.77.2.345. PMID 3276409